CLINICAL TRIAL: NCT06051656
Title: Effect of the Cryoneurolysis on Pain and Positioning in Patients With Wrist and Hand Contractures.
Brief Title: Effect of Cryoneurolysis on Pain in Patients With Hand Contracture.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: H22-03181
Record Dates: First submitted 2023-08-01; First posted 2023-09-25 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Contracture; Spasticity, Muscle
Keywords: Wrist contracture; Severe spasticity; Pain; Cryoneurolysis; Hand contracture
MeSH Terms: conditions — Contracture; Muscle Spasticity; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: Any adult patient with severe hand and wrist spasticity or contracture who suffers from a refractory pain, and is already candidate for cryoneurolysis.

SUMMARY:
Contracture which is defined as a limitation of the maximum passive range of motion due to changes in periarticular soft tissue can contributes to severe pain and increased disabilities. Once contracture is present, management options are very limited and mainly includes surgery. This clinic offers cryoneurolysis routinely to spastic patients to manage their severe spasticity, contracture and associated pain. In this observational project, the outcomes after cryoneurolysis in patients with wrist and hand contracture will be studied systematically and with more details to determine any changes in pain and range of motion after this procedure.

DETAILED DESCRIPTION:
Contracture is defined as a limitation of the maximum passive range of motion of a joint due to shortening and changes of periarticular soft tissue structures. Contracture contributes to severe pain, increased disabilities, decreased functional range of motion and decreased functional range of motion in daily living. The incidence of contracture in first year after has been recorded to be as high as 66%and up to 28% within 3 months after stroke. There are many pharmacological and non pharmacological guidelines available for treatment of contracture and associated pain, including botulinum toxin injection, physiotherapy, stretching and positioning, though; the surgery has been recommended as the most effective one .

Cryoneurolysis is a novel procedure that causes nerve degeneration by cooling them to -88°. The first step in this procedure is isolating the targeted nerves with ultrasound guidance and e-stimulation for motor nerves and mixed sensory motor nerves for pain management. To select the proper candidate for this procedure, targeted nerves will be temporary paralyzed by blocking them with lidocaine (DNB). In this clinic after successful DNB to reduce pain and muscle tone, the patient is offered cryoneurolysis. After rapid cooling the nerve to a certain degree the axon and myelin of targeted zone will be disrupted however ; the basal lamina, epineurium and perineurium of the targeted nerves will be remained intact and serve as a tube for neural regeneration.

This observational study, proposes to measure the effect of cryoneurolysis prospectively and systematically on pain reduction in patients with wrist and hand severe spasticity or contracture due to any underlying disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients(at least 18 years old).
2. Severe claw hand with less than 4 cm distance between the pulp of the fingers and palm of the hand.
3. MAS>= 3 in wrist and hand muscles interfering with function or causing a clinical problem, due to any neurological condition.
4. Have refractory pain in wrist and hand areas with no response to the usual pain management methods including oral medication or botulinum toxin injection.
5. Patients are already candidate for cryoneurolysis to manage the pain and spasticity in their hand and wrist, based on their response to diagnostic nerve block test (DNB).
6. Ability to attend testing sessions, comply with testing protocols and provide written informed consent. For patients who physically are not able to complete the consent process, a witness may be asked to sign and confirm their willing for participation. Legal representative may be asked to help with consent process for participants who cognitively are not able to consent on their behalf.

Exclusion Criteria:

1. Have undergone any previous peripheral nerve procedures in their affected side, for the treatment of spasticity, including previous cryoneurolysis, chemical neurolysis, neurectomy or arthroplasty.
2. Patients who received botulinum toxin in past 4 months in the same targeted muscles for cryoneurolysis, however, they may enter the study at the 4-month mark.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient with wrist/hand contracture and a refractory pain who is already a candidate for cryoneurolysis based on their response to the diagnostic nerve block test (DNB).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Any changes in wrist and hand pain after cryoneurolysis. | The assessment will be done at baseline, 2 weeks, 1 and 4 months after the procedure.
  The intensity of pain in wrist and hand area will be measured based on numerical rating scale (NRS) on scale of 0 to 10 (0 means no pain at all and 10 shows the worst pain that the patient reports).
Any changes in wrist and hand pain after cryoneurolysis , in patients who are not cognitively able to report the intensity of pain. | The assessment will be done at baseline, 2 weeks, 1 and 4 months after the procedure.
  Patients who cognitively are not able to score their pain based on NRS, will be assessed by checklist of nonverbal pain indicators (CNPI). In this scale the patients will be observed in rest and during any movement, and any non verbal or verbal complaints, facial grimaces, bracing, restlessness, rubbing of the affected area will be recorded. The presence or absence of these symptoms will be recorded.
Any changes in wrist and hand spasticity and tone. | The assessment will be done at baseline, 2 weeks, one and four months after the procedure.
  The degree of spasticity will be measured based on Modified Ashworth Scale (MAS) . This scale has 6 scores from 0 which means no spasticity to 4 which means the maximum tone in which the limb movement is limited.
Any changes in wrist and hand range of motion will be recorded. | The assessment will be done at baseline, 2 weeks, one and four months after the procedure.
  Maximum passive and active range of motion of wrist , second and fifth metacarpophalangeal (MCP) and proximal interphalangeal (PIP) joints and thumb radial and palmar abduction will be measured using a goniometer.

SECONDARY OUTCOMES:
Any changes in maximum distance between pulp of the fingers and palm of the hand. | The assessment will be done at baseline, 2 weeks, one and four months after the procedure.
  The maximum distance between the pulp of most flexed finger and palm of the hand will be measured in centimetre. The same measurement will be done for distance between pulp of thumb and palm of the hand.
Any changes in hand hygiene will be recorded. | The assessment will be done at baseline, 2 weeks, one and four months after the procedure.
  Patients' hands will be assessed to determine the extent of any palm maceration, ulceration or infection; cleanliness of the palm, ease of cleaning and nail trimming; and the effect of hygiene-related disabilities on other area of functioning. This assessment is a part of disability assessment scale (DAS). Each section's score ranges from 0 to 3 (0= no disability and 3 = maximum disability)
Patients satisfaction on pre set goals, after the procedure. | The assessment will be done at baseline and at 4 months.
  Goal attainment scale (GAS) is a patient oriented scale to score patients satisfaction with their desired outcomes. Before the procedure up to 3 individualized goals will be negotiated between patients, their caregivers and physicians. At the final visit they will be asked if they are satisfied with each of these goals, and their responses will be scored accordingly. The scores of (-2), (-0.5), (0), (+1) and (+2) will be assigned if they feel that their condition is worse than before, better but not as good as expected, as expected, better than expected and much better than expected. All goals will be weighted equally, and final score will be calculated based on the available formula. The higher score is presenting of better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Paul Winston, MD, Principal Investigator — Vancouver Island Health
Locations (1):
- Victoria General Hospital, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.

REFERENCES:
- [Background] Clavet H, Hebert PC, Fergusson D, Doucette S, Trudel G. Joint contracture following prolonged stay in the intensive care unit. CMAJ. 2008 Mar 11;178(6):691-7. doi: 10.1503/cmaj.071056. PMID 18332384
- [Background] Diong J, Harvey LA, Kwah LK, Eyles J, Ling MJ, Ben M, Herbert RD. Incidence and predictors of contracture after spinal cord injury--a prospective cohort study. Spinal Cord. 2012 Aug;50(8):579-84. doi: 10.1038/sc.2012.25. Epub 2012 Mar 27. PMID 22450888
- [Background] Matozinho CVO, Teixeira-Salmela LF, Samora GAR, Sant'Anna R, Faria CDCM, Scianni A. Incidence and potential predictors of early onset of upper-limb contractures after stroke. Disabil Rehabil. 2021 Mar;43(5):678-684. doi: 10.1080/09638288.2019.1637949. Epub 2019 Jul 22. PMID 31328966
- [Background] Schnitzler A, Diebold A, Parratte B, Tliba L, Genet F, Denormandie P. An alternative treatment for contractures of the elderly institutionalized persons: Microinvasive percutaneous needle tenotomy of the finger flexors. Ann Phys Rehabil Med. 2016 Apr;59(2):83-6. doi: 10.1016/j.rehab.2015.11.005. Epub 2016 Jan 13. PMID 26797076
- [Background] Ilfeld BM, Gabriel RA, Trescot AM. Ultrasound-guided percutaneous cryoneurolysis for treatment of acute pain: could cryoanalgesia replace continuous peripheral nerve blocks? Br J Anaesth. 2017 Oct 1;119(4):703-706. doi: 10.1093/bja/aex142. No abstract available. PMID 29121277

DOCUMENTS (1):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT06051656/Prot_000.pdf